CLINICAL TRIAL: NCT00959517
Title: Pseudo-randomised, Double-blinded Placebo-controlled Trial of Chloroquine or Sulphadoxine-pyrimethamine Alone or in Combination With Primaquine or Artesunate for the Treatment of Uncomplicated Falciparum Malaria in Pakistan
Brief Title: Trial of Artesunate Combination Therapy in Pakistan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: HealthNet TPO (Other)
Responsible Party: Dr Mark Rowland, London School of Hygiene & Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T26/181/33 A00017; TDR A00017
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Uncomplicated Falciparum Malaria
Keywords: Placebo controlled; Efficacy; Artemisinin-based combination therapy; Primaquine; Gametocytes
MeSH Terms: interventions — Artesunate; fanasil, pyrimethamine drug combination; Chloroquine; Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- CQ (Experimental)
  Interventions: Drug: Chloroquine (CQ)
- CQ+PQ (Experimental)
  Interventions: Drug: Chloroquine (CQ); Drug: primaquine (PQ)
- CQ + AS (Experimental)
  Interventions: Drug: artesunate (AS); Drug: Chloroquine (CQ)
- SP (Experimental)
  Interventions: Drug: sulphadoxine-pyrimethamine (SP)
- SP + PQ (Experimental)
  Interventions: Drug: sulphadoxine-pyrimethamine (SP); Drug: primaquine (PQ)
- SP + AS (Experimental)
  Interventions: Drug: artesunate (AS); Drug: sulphadoxine-pyrimethamine (SP)

INTERVENTIONS:
Drug: artesunate (AS) — Recommended dosage over 3 days (for all interventions)
  Arms: CQ + AS; SP + AS
Drug: sulphadoxine-pyrimethamine (SP)
  Arms: SP; SP + AS; SP + PQ
Drug: Chloroquine (CQ)
  Arms: CQ; CQ + AS; CQ+PQ
Drug: primaquine (PQ)
  Arms: CQ+PQ; SP + PQ

SUMMARY:
This study is an evaluation of the benefit of adding artesunate to existing first and second line antimalarial therapies in Pakistan.

A placebo controlled trial was carried out to assess two potential benefits of Artesunate Combination Therapy (ACT): efficacy and potential for transmission reduction.

DETAILED DESCRIPTION:
A randomised, double-blind placebo controlled study of the efficacy of chloroquine or sulphadoxine-pyrimethamine alone and in combination with primaquine or artesunate for the treatment of uncomplicated falciparum malaria.

Arms:

1. CQ
2. CQ+primaquine
3. CQ+ artesunate
4. SP
5. SP+primaquine
6. SP+artesunate

Patients were allocated to treatment groups using a pseudo-randomised table split by age and sex.

Primary outcomes:

* Clinical and parasitological cure/treatment failure by day 28.

Secondary outcomes:

* time to resolution of fever
* time to clearance of trophozoites
* time to clearance of gametocytes
* gametocyte carriage on or after day 7 after treatment

All clinical assessments and slide readings were carried out by staff blind to treatment arm. Slides were double read.

ELIGIBILITY:
Inclusion Criteria:

* presentation at basic health unit with suspected clinical malaria
* mono-infection infection with P. falciparum confirmed by microscopy
* over 2 years of age (no upper age restriction)
* weight over 5 kg (no upper weight restriction)
* if of child bearing age then non-pregnant and willing to remain so for the duration of the study
* greater than 1 asexual parasite per 10 fields
* understands and is willing to sign the consent form
* a resident in the study site willing to collaborate for a full period of follow-up
* no signs of severe malaria

Exclusion Criteria:

* other serious disease (e.g., cardiac, renal or hepatic)
* in women of child bearing age, pregnancy
* allergy to any of the study drugs or related compounds
* reports to have used any malaria drugs in the last 21 days
* other species of malaria seen
* signs of severe malaria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2001-07; Primary Completion 2005-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Parasitological outcome after 28 days follow-up | 28 days

SECONDARY OUTCOMES:
Asexual parasite clearance by day 7 | 7 days
Gametocyte carriage on or after day 7 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Rowland, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- HealthNet International, Peshawar, Pakistan

REFERENCES:
- [Derived] Kolaczinski K, Leslie T, Ali I, Durrani N, Lee S, Barends M, Beshir K, Ord R, Hallett R, Rowland M. Defining Plasmodium falciparum treatment in South West Asia: a randomized trial comparing artesunate or primaquine combined with chloroquine or SP. PLoS One. 2012;7(1):e28957. doi: 10.1371/journal.pone.0028957. Epub 2012 Jan 31. PMID 22303437